CLINICAL TRIAL: NCT01627483
Title: Improving Treatment With Fracture-preventing and Fall-risk-increasing Drugs in Older Hip Fracture Patients: Effects of Medication Reviews Performed by a Physician - a Randomized Controlled Trial
Brief Title: Randomized Controlled Trial of Effects of Physician's Medication Reviews on Prescribing in Older Hip Fracture Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: Ministry of Health and Social Affairs, Sweden (Other Government)
Responsible Party: Principal Investigator, Christina Sjoberg, MD, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SUCPGMHip-09; 095-09 (Other: Regional Ethical Review Board in Gothenburg)
Record Dates: First submitted 2012-06-21; First posted 2012-06-25 (Estimated); Last update posted 2012-06-25 (Estimated); Status verified 2012-06

CONDITIONS: Hip Fracture
Keywords: elderly; hip fracture; osteoporosis; fall risk; medication review
MeSH Terms: conditions — Hip Fractures; Osteoporosis | interventions — Medication Review

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Medication review (Experimental): Assessment of risks of falls and fractures, medication review
  Interventions: Other: Medication review
- Controll (No Intervention)
  Interventions: Other: Medication review

INTERVENTIONS:
Other: Medication review — Assessment of risks of falls and fractures; medication review concerning fall-risk-increasing and fracture-preventing drugs; oral and written feed back of the results of the assessments and medication reviews to the hospital physician during the hospital stay and to the general practitioner 3 and 6 months after the hip fracture surgery.

SUMMARY:
The aim of this study is to investigate if prescribing of fall-risk increasing and fracture-preventing drugs can be improved in older hip fracture patients by assessments of risks of falls and fractures and medication reviews performed by a physician and forwarded to prescribing physicians.

DETAILED DESCRIPTION:
The patients will be recruited postsurgery. They will be randomly allocated to an intervention or a control group (1:1). Sequentially numbered, opaque, sealed envelopes will be opened sequentially after participant details are written on the envelope. Carbon paper inside the envelope will transfer the information to the assignment card. Two persons not involved in the study and without knowledge about the study protocol will perform the randomization procedure. The patient will not be informed about the result of randomization.

Intervention By a short interview and/or extraction of information from the medical records comprehensive assessments of the risk of falls and the risk of fractures. Thereafter a medication review focusing on fall-risk-increasing and fracture-preventing drugs will be performed. The results of the assessments and the medication review will be forwarded orally and in written to the prescribing physicians. The recipients will be the physician at the ward during inhospital care and the general practitioner at three and six months after the surgery.

Data collection Prescribing of drugs Data will be obtained from the medical records of Sahlgrenska University Hospital, the medical records of the general practitioner, the multi-dose drug dispensing list, if any, and the Swedish Prescribed Drugs Register (Läkemedelsförteckningen).

Patient data Information on the patients during the hospital stay and the follow-up period will be obtained from the medical records of the hospital, the medical records of the general practitioner, the Swedish National Hip Fracture Register (RIKSHÖFT), and from the health care database in the Region of Västra Götaland. Data on other medical care contacts due to a fall accident will be obtained from the care database in the Western Region (VEGA database). Additionally, data on diagnoses will be obtained from the National Patient Register (Patientregistret). For deceased patients, data from the Cause of Death Register (Dödsorsaksregistret) will be obtained.

Physicians attitudes A short questionnaire will be administered to the physicians at the hospital and the general practitioners. The questionnaire will be answered anonymously and will include questions on attitudes towards the intervention and its usefulness. A reminder will be administered two weeks later.

Power calculation The study has a power of >80% to detect a 50% rise in the prescribing of fracture-preventing drugs in the intervention group, a doubling in bisphosphonates or other bone specific drugs and a reduction of 15% in the mean (SD) number of fall-risk increasing drugs. Power calculations were based on the assumption that drug treatment in the control group was improved by 30% for all fracture-preventing drugs and 60% for bisphosphonates when compared with the study performed in 2008.

ELIGIBILITY:
Inclusion Criteria:

* hip fracture surgery at Sahlgrenska University Hospital/Mölndal
* aged 65 years and over
* residing in the Gothenburg area

Exclusion Criteria:

* own opposition to participation
* if not able to give informed consent, opposition to participation by next of kin

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Actual)
Dates: Start 2009-04; Primary Completion 2010-04 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Treatment with fall-risk-increasing drugs | One year
  Drug treatment is estimated from the Swedish Register of Dispensed Drugs
Treatment with fracture-preventing drugs | One year
  Drug treatment is estimated from the Swedish Register of Dispensed Drugs

SECONDARY OUTCOMES:
Attitudes towards the intervention among physicians | Ten months
  Attitudes towards the oral and written parts of the intervention are investigated by a short questionnaire sent to the involved physicians and answered anonymously.
Fall-related injuries in need of medical care | One year
  Contact with a physician due to an injury caused by a fall
Death | One year

CONTACTS AND LOCATIONS:
Overall Officials: Susanna M Wallerstedt, Assprofessor, Study Director — Department of Clinical Pharmacology, Sahlgrenska University Hospital, Bruna stråket 21, S-413 45 Gothenburg, Sweden
Locations (1):
- Sahlgrenska University Hospital/Mölndal, Mölndal, Region Västra Götaland, Sweden

REFERENCES:
- [Background] Sjoberg C, Bladh L, Klintberg L, Mellstrom D, Ohlsson C, Wallerstedt SM. Treatment with fall-risk-increasing and fracture-preventing drugs before and after a hip fracture: an observational study. Drugs Aging. 2010 Aug 1;27(8):653-61. doi: 10.2165/11538200-000000000-00000. PMID 20658793